CLINICAL TRIAL: NCT03739086
Title: Evaluation of Erector Spinae Plane Block; Indications, Complications and Analgesic Effects
Brief Title: Retrospective Evaluation of Erector Spinae Plane Blocks
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., assoc professor in anesthesiology department, Maltepe University
Other Study IDs: ESPB-retro
Record Dates: First submitted 2018-10-21; First posted 2018-11-13 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: erector spinae plane block — unilateral or bilateral or bilevel erector spinae plane block performance for postoperative pain or acute pain

SUMMARY:
Retrospective Evaluation of Erector Spinae Plane Blocks

DETAILED DESCRIPTION:
in our institue; we use erector spinae plane block as a part of multimodal analjesia. we want to evaluate block failures and complications related erector spinae plane block. In all patients performed regional anesthesia techniques, we use a regional anesthesia follow chart.

ELIGIBILITY:
Inclusion Criteria:

* patient performed erector spinae plane block

Exclusion Criteria:

-

Max Age: 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all of the patients performed erector spinae plaen block
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
complication rate | 14 months

SECONDARY OUTCOMES:
block failure rate | 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Result] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005